CLINICAL TRIAL: NCT03560713
Title: Effects of Functional Electrical Stimulation in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Isabella Martins de Albuquerque, Professor DSc, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 85774518.3.0000.5346
Record Dates: First submitted 2018-05-24; First posted 2018-06-18 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Muscle Wasting
MeSH Terms: conditions — Muscular Atrophy | interventions — proto-oncogene protein c-fes-fps; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES + combined exercise (Experimental): The Functional Electrical Stimulation (FES) + combined exercise group will receive 12 weeks of FES (Neurodyn High Volt, IBRAMED, São Paulo/SP, Brasil), three times a week, frequency 25Hz, pulse rate of 200μs, ON:OFF 5:5, individual maximum tolerated intensity; minimum at strong but comfortable visible muscle contraction (without causing undue pain or discomfort to the participant) and receive aerobic exercise training and resistance exercises for upper limbs and lower limbs.
  Interventions: Device: Functional Electrical Stimulation (FES)
- FES sham (Sham Comparator): The Functional Electrical Stimulation (FES) sham + combined exercise group will receive 12 weeks of FES (Neurodyn High Volt, IBRAMED, São Paulo/SP, Brasil), three times a week, frequency 5Hz, pulse rate of 200μs, ON:OFF 5:5, without muscle contraction during 30 minutes and receive aerobic exercise training and resistance exercises for upper limbs and lower limbs.
  Interventions: Other: Functional Electrical Stimulation (FES) sham

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) — Participants will perform 12 weeks of FES (Neurodyn High Volt, IBRAMED, São Paulo/SP, Brasil), three times a week, frequency 25Hz, pulse rate of 200μs, ON:OFF 5:5, individual maximum tolerated intensity; minimum at strong but comfortable visible muscle contraction (without causing undue pain or discomfort to the participant). during 30 minutes nd receive aerobic exercise training and resistance exercises for upper limbs and lower limbs.
  Other Names: FES + combined exercise
  Arms: FES + combined exercise
Other: Functional Electrical Stimulation (FES) sham — Participants will perform 12 weeks of Functional Electrical Stimulation (FES) sham (Neurodyn High Volt, IBRAMED, São Paulo/SP, Brasil), three times a week, frequency 5Hz, pulse rate of 200μs, ON:OFF 5:5, without muscle contraction during 30 minutes nd receive aerobic exercise training and resistance exercises for upper limbs and lower limbs.
  Other Names: FES sham + combined exercise
  Arms: FES sham

SUMMARY:
Even with major advances in clinical therapy and percutaneous interventions, coronary artery bypass grafting (CABG) is the most common cardiac surgery performed worldwide and is an effective treatment in reducing symptoms and mortality in patients with coronary artery disease (CAD). However, CABG is a complex procedure that triggers a series of clinical and functional complications, such as series postoperative repercussions as muscle wasting in the first four hours after surgery. For quantification of changes in muscle structure and morphology ultrasonography has been used.

In this context, cardiac rehabilitation program (CRP) is an essential component of care in CABG patients, because this intervention can prevent muscle weakness and wasting. Among different treatment modalities, functional electrical stimulation (FES) is a feasible therapy for neuromuscular activation and prevent muscle weakness and wasting in patients in phase I CRP, however the effect of this intervention in phase II CRP not been fully elucidated. The purpose of this study will to assess the effects of FES plus combined aerobic and resistance training on muscle thickness of quadriceps femoris, lower limbs muscle strength, functional capacity, QoL in in CABG patients enrolled in a phase II CR program.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing CABG up to three weeks before the initiation of the study, a clinical course without complications during hospitalization

* Clinically stable
* The absence of smoking (previous or current).

Exclusion Criteria:

* Unstable angina
* Myocardial infarction and heart surgery up to three months before the survey
* Chronic respiratory diseases
* Hemodynamic instability
* Orthopedic and neurological diseases that may preclude the achievement of the cardiopulmonary test and Cardiac Rehabilitation exercises
* Psychological and/or cognitive impairment that restrict them to respond to questionnaires
* Changes of skin sensitivity,skin lesion and allergic skin problems
* Severe lymphedema
* Uncontrolled diabetes mellitus
* Acute superficial venous thrombophlebitis
* Systemic arterial hypertension

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Muscle thickness of the quadriceps femoris | Change in muscle thickness (in cm) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Muscle thickness of the quadriceps femoris will be assessed by ultrasonography (baseline and after 12 weeks)

SECONDARY OUTCOMES:
Vastus intermedius, rectus femoris echo intensity | Change in vastus intermedius and rectus femoris echo intensity (in region of interest -ROI) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Vastus intermedius, rectus femoris echo intensity will be assessed by ultrasonography (baseline and after 12 weeks)
Rectus femoris cross-sectional area | Change in rectus femoris cross-sectional area (in cm2) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Rectus femoris cross-sectional area will be assessed by ultrasonography
Rectus femoris and vastus intermedius thickness | Change in rectus femoris and vastus intermedius thickness (in cm) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Rectus femoris and vastus intermedius thickness will be assessed by ultrasonography
Ankle-brachial index | Change in ankle-brachial index (in mmHg) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Ankle-brachial index will be assessed by by Doppler ultrasonography using color Doppler.
Peripheral muscle strength of the lower limbs | Change in peripheral muscle strength (in number of repetitions performed in the STST) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Peripheral muscle strength of the lower limbs will be measured by sit-to-stand test (STST).
Peripheral muscle strength of the lower limbs | Change in peripheral muscle strength (in the maximum load (kg) lifted up during the one-repetition maximum test ) from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Peripheral muscle strength of the lower limbs will be measured by one-repetition maximum muscle strength.
Quality of life | Change in MacNew scores from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Quality of life will be measured by a MacNew Heart Disease health-related quality of life instrument
Lower-limb functional exercise capacity | Change in distance walked (meters) by the patients during six-minute walk test from baseline at after 12 weeks of rehabilitation cardiac admission, an average of 3 months
  Lower-limb functional exercise capacity will be assessed by six-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Isabella Martins de Albuquerque, Santa Maria, Rio Grande do Sul, Brazil